# Prevent Cardiac Surgery Associated Acute Kidney Injury Trial (Prevent CSA-AKI Trial)

Efficacy of Mitochondrial directed therapy in prevention of cardiac surgery associated acute kidney injury

NCR224635 Data Dictionary

19-Feb-2024

# A -Demographics

- 1- Date of admission
- 2- Surgery start date/time
- 3- Surgery end date/time
- 4- ICU admission date/time
- 5- ICU discharge date/time
- 6- Hospital discharge date/time
- 7- Hospital discharge date/time
- 8- Readmission to ICU date #1
- 9- Readmission to ICU date #2
- 10-Readmission to ICU date #3
- 11-Age on admission
- 12-Sex
  - a. Male
  - b. Female
- 13-Weight on admission
- 14-Race
  - a. Asian
  - b. Black
  - c. White
  - d. American Indian or Alaska Native
  - e. Native Hawaiian or Another Pacific Islander
  - f. Other
- 15-Ethnicity
  - a. Hispanic
  - b. Non-Hispanic
- 16-BMI on admission
- 17-H/o of cancer (type)
  - a. Free text
- 18-H/o of systolic heart failure (options below)
  - a. Acute
  - b. Chronic
  - c. Acute on chronic
- 19-H/o of diastolic heart failure (options below)
  - a. Acute
  - b. Chronic
  - c. Acute on chronic
- 20-History of combined HF (systolic and diastolic) (18 and 19 cannot be yes if 20 is yes)
- 21-EF (%)
- 22-History of CAD

### 23-Valvular heart disease (valve)

- a. Aortic Valve disease
- b. Mitral Valve disease
- c. Tricuspid Valve disease
- d. Pulmonic Valve disease

#### 24-COPD

### 25-DM

- a. Type I
- b. Type II

#### **26-HTN**

- 27-CKD stage III A
- 28-H/o of Atrial fibrillation
- 29-H/o Stroke
- 30-H/o of hypothyroidism
- 31-H/o of liver Cirrhosis
- 32-H/o of transplant (type free text)
- 33-Immunosuppression
- 34-H/o of autoimmune disease
- 35-H/o of HIV

## B- Surgery & Cardiac devices :

## 1-Typer of surgery :

- Single valve
- >1 valve
- CABG
- Combined CABG and ≥ 1 valve
- Other

### 2-Cardiopulmonary bypass details:

- Skin incision start date/time
- Skin incision stop date/time
- Aortic cross clamp time (minutes)
- Cardio Pulmonary Bypass time (minutes)
- Lowest hematocrit % recorded in the OR
- Episode of MAP <50
- Episode of MAP < 50 for > 15 consecutive minutes

### 3- Cardiac devices (start and stop):

- Impella (2.5 Vs 5)
- IABP
- ECMO (VA vs VV vs VAV)
- LVAD

## C- New Diagnosis during admission:

- New A fib
- ≥ 2 Sustained V tach episodes
- Bradycardia
- Complete heart block
- Cardiac arrest
- New pacemaker
- Pericarditis
- Pericardial effusion
- EF (changes in EF %)
- Cardiac tamponade
- Stroke
  - Hemorrhagic/location (free text for location)
  - Embolic/territory (free text for territory)
- Perioperative MI
- Graft occlusion
- Sepsis & source (yes/no; free text for source)
- Return to OR #1
  - Date
  - Reason (free text)
- Return to OR #2
  - Date
  - Reason (free text)
- Return to OR #3
  - o Date
  - Reason (free text)
- Return to OR #4
  - o Date
  - Reason (free text)
- Return to OR #5
  - o Date
  - Reason (free text)
- Presence of bacteremia (source)
- Digit ischemia
- Intestinal /bowel/mesenteric ischemia
- Bleeding (location as free text)

## D - Home Medications (all as yes/no)

- ACE I & ARB: Lisinopril, Enalapril, Captopril, Iosartan, Valsartan, Entresto
- Other Anti hypertensives: amlodipine, nifedipine, hydralazine, clonidine, imdur, doxazosine
- SGLT inhibitors: Empagliflozin, dapagliflozin, canagliflozin, ertugliflozin
- MRA: Spironolactone, Eplerenone
- Diuertics: hydrochlorothiazide, furosemide, Torsemide, bumetanide, metolazone, chlorothiazide
- Betablockers : Sotalol Labetalol Metoprolol. Atenolol Bisoprolol Carvedilol, Nadolol Nebivolol
- Other AV node blocker: Amiodarone Digoxin, Diltiazem, Disopyramide, Dofetilide, Dronedarone, Flecainide, Propafenone, Quinidine sulfate, Verapamil

# **E-ICU medications** (start and stop dates of the meds below, repeat entry as needed only if stopped ≥ 1 day)

- Pressor (Epi, NE, Neo, Vaso, ATII)
- Milrinone
- Dobutamine
- Diuertics: hydrochlorothiazide, furosemide, Torsemide, bumetanide, metolazone, chlorothiazide, spironolactone, eplerenone
- Hypertension meds: Amlodipine, nifedipine, hydralazine, clonidine, imdur, doxazosin
- BB: Sotalol, Labetalol, Metoprolol, Atenolol, Bisoprolol, Carvedilol, Nebivolol
- ACE I & ARB : Lisinopril, Enalapril, Captopril, Iosartan, Valsartan, Entresto
- SGLT inhibitors: Empagliflozin, dapagliflozin, canagliflozin, ertugliflozin)
- Other AV node blocker: Amiodarone, Digoxin, Diltiazem, Verapamil
- Dexmedetomidine

## F. General Labs:

One set prior to OR and daily during admission if availble

- (Hemoglobin, Hematocrit, WBC, Platelets, BUN, Creatinine, eGFR, Bicarbonate, ALT, AST, bilirubin, Albumin, Magnesium, Potassium, sodium, Blood sugar, calcium, BNP, TSH, trop, lactic acid, INR.
- ABG (Ph, Pco2, Po2, Fio2)
- UA: proteinuria
- Urine protein creatinine ratio
- Urine albumin

# G. Special labs (NIH):

- Serum and urinary levels of CoQ10, glutathione, serum and Urinary mtDNA

1<sup>st</sup> samples in the week prior to surgery

2<sup>nd</sup> sample in Day 0; the day of surgery

3<sup>rd</sup> sample in Day 1; the day after surgery

### H. Clinical

### 1-Vitals:

- Prior to surgery: Heart rate, MAP, saturation
- Recording daily MAP, HR, Sat: (Mode: most common number for the day)
  - Number of Episodes of MAP <50</li>
  - o Number of episode of MAP < 50 for > 15 consecutive minutes
- **2- Respiratory:** level of support daily including day prior to surgery (report only the final modality and amount of O2 support for each day)
- RA
- Nasal cannula
- HFNC
- BiPAP/ CPAP
- Vent
  - Mode
  - o PEEP
  - o Fio2
  - $\circ$  RR
  - o start and stop date

# 3-Renal Replacement Therapy (RRT)

- CRRT (CVVH or CVVHD), start date, stop date
- Hemodialysis start and stop date

### 4- Volume status:

Daily Ins Daily out Daily Chest tube drainage Daily urine output

### 5-Adverse events:

- Nausea
- Vomiting
- Diarrhea
- Rash
- Loss of appetite
- Other (free text)

# I- evaluations/ calculations within 28 & 90 days:

- Apache & Sofa score calculation during ICU stay
- AKI stage
- AKD and CKD
- RRT dependence
- RRT free days
- Ventilator free days
- Death
- MAKE within 30 & 90 days
- Readmission (number/ dates/ reasons)

## J. Definitions:

- AKI is defined as 2012 KDIGO guideline •Increase in SCr by equal or more than 0.3 mg per dl (equal or more than 26.5 µmol per l) within 48 hours; or •Increase in SCr to equal or more than 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or •Urine volume less than 0.5 ml per kg per h for 6 hours
- RRT dependence defined by the receipt of any form of RRT within + or 14 days of the 90- day time point following randomization.
- RRT free days as the number of days between s from RRT and day 28 after study

Ventilator free days as the number of days between successful weaning from mechanical ventilation and day 28 after study enrollment

- Ventilator-free day is defined as the receipt of less than 2 hours of invasive or noninvasive ventilation within a 24-hour period.
- Shock-free days defined as less than 2 hours of receipt of any vasoactive therapy provided by continuous infusion within a 24-hour period.
- -Make within 30 & 90 days ( major adverse kidney events ) defined by 1 or more of the following:
  - In hospital mortality
  - Death prior to discharge
  - New receipt of RRT (any modality prior to hospital discharge)

Persistent renal dysfunction (final Creatinine before discharge ≥ 200% of the baseline Cr value in a patient not know to have previously received RRT

